CLINICAL TRIAL: NCT03842280
Title: Assessments of Diaphragm-pleural Mechanics During the Weaning From Prolonged Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201811015RINA
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Ventilator Weaning; Respiratory Failure
Keywords: Prolonged mechanical ventilation; Esophageal pressure; Pleural pressure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prolonged mechanical ventilation: Prolonged mechanical ventilation with tracheostomy
  Interventions: Device: Diaphragm ultrasound assessment & Esophageal pressure measurement

INTERVENTIONS:
Device: Diaphragm ultrasound assessment & Esophageal pressure measurement — Diaphragm ultrasound assessment and/or Esophageal pressure measurement before, during and after spontaneous breathing trial

SUMMARY:
Weaning failure from mechanical ventilator is commonly seen in respiratory failure and increases duration of ventilator use, ICU stay, ventilator associated pneumonia and even mortality. The diaphragm serves as one of the most important respiratory mechanism and its function differs the weaning success rate. Since 1980s, ultrasonography assessment in diaphragm movement were developed and further discussion upon whether it serves as a predicting factor for extubation failure. The measurement includes difference of diaphragm thickness, diaphragm excursion or the movement of liver and spleen.

Multiple studies targeted intubated patients with different measurement methods and all resulted with good weaning prediction value.6 Of all the studies, only one study targeted tracheostomy tube patients. They reported diaphragm thickness fraction >36% as cutoff value is associated with successful spontaneous breathing trial (SBT), with a sensitivity of 0.82, specificity of 0.88. However, little comparison with traditional weaning parameters was mentioned in the study. We designed this prospective observational study to evaluate whether diaphragm movement under ultrasound serves as a predicting index of ventilator discontinuation in patients with tracheostomy. The diaphragm movement will also correlate with other parameters such as RSBI, Pi max, Pe max, Tv spont., WEANSNOW score(WS), VO2, APACHE II. Esophageal pressure is also provided as an option for our study population for more information such as pleural pressure, transdiaphragm pressure, etc.

The ultrasonography measurement of diaphragm movement will be performed within 6 hours before discontinuation of ventilator. The patient remains in semi-recumbent position with the convex probe selected for its good penetration. The probe is placed at a craniocaudal axis, 90 degrees to the skin at the lower intercostal spaces to right anterior axillary line (AAL) and left posterior axillary line (PAL), which allows a perpendicular ultrasound beam direction to the diaphragm movement. Liver (border or vascular structure), splenic (border or vascular structure) will be selected as target point and the marked distance of movement during quiet respiration cycle will be measured 10 times with a largest value calculated. Other echo measurements will also be attempted.

The study aims to investigate if the measurement of the diaphragm movement serves as a reliable predicting factor for weaning failure in respiratory care center patients.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged mechanical ventilation with tracheostomy tube
* Oxygen with a fraction of ≤ 0.4
* Positive end expiratory pressure at ≤ 5 cm H2O
* Pressure support at ≤ 8 cmH2O

Exclusion Criteria:

* No spontaneous breathing
* Unstable hemodynamic status,
* History of peritonitis, intraabdominal operation, empyema, or pleurodesis.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with prolonged mechanical ventilation with tracheostomy tube with admission to respiratory care center in NTUH
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Weaning success | 1 month
  Liberation from mechanical ventilation

SECONDARY OUTCOMES:
Ventilator free 30 days after liberation | 30 days after liberation
  No mechanical ventilation use in 30 days after liberation
Ventilator free 60 days after liberation | 60 days after liberation
  No mechanical ventilation use in 30 days after liberation
Ventilator free 90 days after liberation | 90 days after liberation
  No mechanical ventilation use in 90 days after liberation

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan